CLINICAL TRIAL: NCT00965679
Title: X-ray Fluoroscopy Fused With Computed Tomography (XFC) Technical Development
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090211; 09-H-0211
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-05-27

CONDITIONS: Aortic Valve Stenosis
Keywords: Cardiac CT; Iodinated Radiocontrast; Ionizing Radiation; Aortic Valve Stenosis; Percutaneous Aortic Valve Replacement; Heart Valve
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* Computed tomography (CT) creates three-dimensional images based on X-ray imaging. CT is useful for determining treatment approaches for certain diseases, such as calcific aortic stenosis (narrowing of the aorta because of calcium deposits).
* Comparing the data received from CT scans with the data received from heart catheterization (which assesses the heart's condition and function) can be used to improve treatment in patients with certain heart conditions. Researchers are interested in looking at the effectiveness of both procedures in assessing possible surgical treatments for patients with calcific aortic stenosis.

Objectives:

- To analyze cardiac CT scans in conjunction with existing heart scan results to improve treatments for future minimally invasive aortic valve replacement.

Eligibility:

- Patients 18 years of age and older who have been diagnosed with aortic valve stenosis that may be treated surgically, and who will undergo or have recently undergone heart catheterization.

Design:

* Participants will have a CT scan within 90 days of the medically necessary heart catheterization, but before any other surgical or catheter treatment.
* During the CT scan, patients will be asked to hold their breath intermittently for about 5 to 20 seconds. Patients will be inside the scanner for less than 30 minutes.
* Patients will be asked to return in 3 to 7 days for a blood test to check kidney function.
* Researchers will analyze the results of the CT scan in conjunction with the previous results from the catheterization to determine possible improved treatment options.

DETAILED DESCRIPTION:
We will collect cardiac computed tomography (CT) data from patients with aortic valve stenosis being considered for surgical or catheter treatment. These data will be analyzed along with medically-necessary fluoroscopy from cardiac catheterization to learn whether they can be combined to enhance future minimally invasive valve treatments.

ELIGIBILITY:
* INCLUSION CRITERIA:

SELECTION CRITERIA: PATHWAY FOR RESEARCH CT:

* Adult patients age 18 years or older
* Having calcific aortic stenosis being considered for surgical or catheter-based treatment, determined on physical examination or noninvasive imaging such as echocardiography
* Undergoing diagnostic cardiac catheterization within 1 year
* Able to provide informed consent

ALTERNATIVE SELECTION CRITERIA: PATHWAY FOR ANALYSIS OF MEDICAL DATA:

* Adult patients age 18 years or older
* Having calcific aortic stenosis being considered for surgical or catheter-based treatment, determined on physical examination or noninvasive imaging such as echocardiography
* Undergoing diagnostic cardiac catheterization within 1 year
* Having undergone cardiac CT for medical indications meeting the technical requirements of this protocol
* Able to provide informed consent

EXCLUSION CRITERIA:

SELECTION CRITERIA: PATHWAY FOR RESEARCH CT:

* Pregnant or lactating women
* Decompensated heart failure (unable to lie flat during CT)

EXCLUSION CRITERIA FOR BETA ADRENERGIC BLOCKERS:

* Advanced atrioventricular block (Mobitz Type II second degree or third degree atrioventricular heart block)
* Asthma or chronic obstructive pulmonary disease (emphysema) currently treated with beta adrenergic agonists

EXCLUSION CRITERIA FOR IODINATED RADIOCONTRAST:

-Severe kidney disease (MDRD estimated Glomerular Filtration Rate

< 30mL/min/l.73m(2)).

-Request of referring physician or surgeon not to administer iodinated radiocontrast

ALTERNATIVE SELECTION CRITERIA: PATHWAY FOR ANALYSIS OF MEDICAL DATA:

-None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-08-06; Study Completion 2010-05-27

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gutierrez LF, Silva Rd, Ozturk C, Sonmez M, Stine AM, Raval AN, Raman VK, Sachdev V, Aviles RJ, Waclawiw MA, McVeigh ER, Lederman RJ. Technology preview: X-ray fused with magnetic resonance during invasive cardiovascular procedures. Catheter Cardiovasc Interv. 2007 Nov 15;70(6):773-82. doi: 10.1002/ccd.21352. PMID 18022851
- [Background] Phan A, Dalle S, Thomas L. [Acquired pigmented lesion of the finger pulp]. Ann Dermatol Venereol. 2009 May;136(5):477-8. doi: 10.1016/j.annder.2008.09.020. Epub 2009 Mar 10. No abstract available. French. PMID 19442811
- [Background] Tenaza RR. Songs, choruses and countersinging of Kloss' gibbons (Hylobates klossii) in Siberut Island, Indonesia. Z Tierpsychol. 1976 Jan;40(1):37-52. doi: 10.1111/j.1439-0310.1976.tb00924.x. PMID 1274481